CLINICAL TRIAL: NCT04915742
Title: Master Physiotherapist
Brief Title: The Effect of Group Exercise and Thetahealing on Pain and Quality of Life in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Naciye Dilruba Tektas Gulbil, physioterapist, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/1366
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Fibromyalgia
Keywords: fibromiyalgia; thetahealing; exercises
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomize
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercises and thetahealing (Experimental)
  Interventions: Behavioral: thetahealing and exercises
- exercises (Active Comparator)
  Interventions: Behavioral: exercises

INTERVENTIONS:
Behavioral: exercises — The exercise group ha in FTAs 2, each session will be 30 minutes of evil sown in stretching , which made combining relaxation and strengthening exercises therapeutic exercise program for 6 weeks from the online platform will be implemented in the form of group exercise form is planned.
  Arms: exercises
Behavioral: thetahealing and exercises — The exercise group ha in FTAs 2, each session will be 30 minutes of evil sown in stretching , which made combining relaxation and strengthening exercises therapeutic exercise program for 6 weeks from the online platform will be implemented in the form of group exercise form is planned.
  The exercise and Thetahealing treatment group, on the other hand, is planned for 6 weeks , 1 session per week, 30 minutes per session, in addition to the exercise sessions, the first and last sessions to be individual and personalized .
  Applications will be carried out on the online platform.
  Arms: exercises and thetahealing

SUMMARY:
Summary

Purpose: Determining the Effect of Therapeutic Exercise and Thetahealing on Pain and Quality of Life in Patients with Fibromyalgia Methods: Between February and April 2021, the study started with 58 people who wanted to participate in the study from online platforms and the study was completed with 34 people.

Findings: According to the power analysis, at least 34 people will participate in the study. Participants will be divided into 2 groups as experimental and control, thetahealing and exercise will be applied to the experimental group and only exercise sessions will be applied to the control group. The study will be 2 sessions of online group exercises per week for 6 weeks and 1 session of tehetahealing will be applied to the experimental group for 6 weeks. The evaluation will be carried out in the first week before the sessions start and in the last week after the sessions are completed in the form of an online survey.Summary

Purpose: Determining the Effect of Therapeutic Exercise and Thetahealing on Pain and Quality of Life in Patients with Fibromyalgia Methods: Between February and April 2021, the study started with 58 people who wanted to participate in the study from online platforms and the study was completed with 34 people.

Findings: According to the power analysis, at least 34 people will participate in the study. Participants will be divided into 2 groups as experimental and control, thetahealing and exercise will be applied to the experimental group and only exercise sessions will be applied to the control group. The study will be 2 sessions of online group exercises per week for 6 weeks and 1 session of tehetahealing will be applied to the experimental group for 6 weeks. The evaluation will be carried out in the first week before the sessions start and in the last week after the sessions are completed in the form of an online survey.

DETAILED DESCRIPTION:
Login Fibromyalgia (FM) is a non-articular, chronic rheumatic disease of unknown etiology, characterized by widespread musculoskeletal pain, sleep disturbance, fatigue, and the presence of multiple tender points (1). Diagnostic criteria were defined by the American Rheumatism Association (ARA) in 1990 (2). In order to diagnose FM, there should be widespread pain and sensitivity in 11 or more of 18 specific points (3). The etiopathogenesis of FM is still unknown, but factors such as physical trauma, surgical intervention, infections, acute or chronic emotional stress may play a triggering role (4). Various findings such as muscular symptoms, cognitive complaints, depression, insomnia and fatigue accompanying chronic pain have been described in patients with FM (5). Various psychopathological disorders have been reported in FM. It is estimated that 1/3 of his patients have minor depression or anxiety. However, it is not known whether anxiety and depression in FM cause chronic pain or contribute to the severity of symptoms (3). Despite the various complaints of patients with fibromyalgia, the fact that no significant impairment was found in physical examination and laboratory tests suggests that the symptoms may be psychologically induced (6). Since the etiology of fibromyalgia syndrome is unknown, pharmacological and non-pharmacological treatment methods should be used in patient-specific combinations according to the prominent symptoms and their severity (6).

Mental health as well as the physical health of FMS patients is frequently investigated. It has been observed that depressions accompany FMS in the majority of patients (7 -11). Likewise, FMS patients frequently get various psychiatric comorbidities such as panic disorder and anxiety (12,13). In addition, studies consistently point to an increased rate of designed suicide after the development of fibromyalgia in this patient group due to the burden of the disease and the high prevalence of depression (14-16).

The role of psychological factors in fibromyalgia is a controversial issue. However, many studies have shown that these patients experience deterioration in personality patterns, increased stress levels, anxiety, depression, or other psychological symptoms (17,18). Although psychological factors are not considered to be the primary cause of fibromyalgia, there are findings that depression is a very important predictor of the development of FMS (12,19). On the other hand, researchers have pointed out that fibromyalgia and depression generally have two-way relationships by overlapping (18,20).

Theta gets its name from Teta brain waves. Generally, at night, while sleeping, during deep meditation , and experiencing oneness in the universe, situations occur at the theta wavelength. So the Theta state is a very deep state of relaxation . While in this wavelength , we can easily connect with the brain so that our haunted beliefs here can be controlled. This condition is associated with strong theta rhythmic activity patterns. Theta activities occur in the electroencephalogram (EEG) between the client and the practitioner at a wavelength of 4-7 Hz (21). ThetaHealing® (Vianna Stibal, Kalispell, MT) is a spiritual healing method in which practitioner and client participate in joint meditations during several subliminal sessions. Thetahealing is practiced by people who are internationally trained in this field. It is claimed that these meditation periods are characterized by a "theta state" in which the presence of theta waves in the electroencephalograph (EEG) frequency spectrum of both the practitioner and the client is assumed (21) .

Located above the psychological and physiological bases for fibromyalgia origin information in light of the Fibromyalgia Patients Group Exercise ii and Thetahealing Pain and e on quality of life TKİ designed this study to determine n.

Method Our research is planned to be conducted entirely on an online platform in order not to risk the participants due to the Covid-19 measures. The study will be carried out on a voluntary basis.

Inclusion criteria for the study:

Being between the ages of 18-60 who have previously been diagnosed with fibromyalgia

Symptoms last longer than 3 months

The volunteer's acceptance of participation in the treatment that will continue 2 days a week for 6 weeks ,

Exclusion criteria from the study:

Using psychotropic medication in the last month

Known central or peripheral nervous system disease, progressive neurological damage,

Any serious cardiovascular pathology.

Any musculoskeletal disease other than fibromyalgia,

Presence of uncontrolled hypertension,

Exclusion criteria:

Volunteer's request to leave

Failure to continue training sessions

S studies due to medical treatment received FMS Residence predicting the likelihood of any changes mei

The data of our study will be analyzed with the SPSS (version 22.0) computer program. Descriptive statistics techniques will be used to reveal the averages of all values of the data obtained in the research (percentage and descriptive statistics, mean and standard deviation values , t test, nonparametric tests if necessary ).

Since it will be a volunteer-based study, the volunteer can leave the study at any time.

Evaluation parameters to be used in research:

The socio-demographic information of the individuals who agreed to participate in the study will be obtained.

It will be used 2 times, with all evaluation parameters before and after treatment.

Pg-36 will be used to evaluate the quality of life of the participants, the numerical pain scale will be used to evaluate the pain levels, and the fibromyalgia impact questionnaire will be used to evaluate the effect level of the disease.

Volunteers participating in our study will be randomly divided into 2 groups. In the randomization of the groups, the assignment to the groups will be made with the randomizer program using a computer. R astgel created in one of two exercise group (control group), the other is exercise additional thetahealig (experimental group) group will have.

Thetahealing will be administered by the researcher who is an internationally trained specialist physiotherapist (Appendix 1 Certificate).

The exercise group ha in FTAs 2, each session will be 30 minutes of evil sown in stretching , which made combining relaxation and strengthening exercises therapeutic exercise program for 6 weeks from the online platform will be implemented in the form of group exercise form is planned.

The exercise and Thetahealing treatment group, on the other hand, is planned for 6 weeks , 1 session per week, 30 minutes per session, in addition to the exercise sessions, the first and last sessions to be individual and personalized .

Applications will be carried out on the online platform.

Evaluation methods to be used in the study

Fibromyalgia Impact Questionnaire:

This scale; It measures 10 different characteristics: physical function, feeling unwell, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. Except for the sense of well-being, lower scores indicate improvement or less affected by the disease. FEA is filled by the patient. The maximum possible score for each subtitle is 10. Thus, the total maximum score is 100. While an average FM patient scores 50, more severely affected FM patients usually score above 70 (1).

Short Form-36: SF-36 was developed to evaluate the quality of life. Its validity and reliability study has been carried out in Turkey. SF-36 is used to compare general and specific populations, to demonstrate the health benefits of different treatments, and to monitor patients. The last 4 weeks are taken into account in the evaluation of SF-36, which consists of 36 items ( 2-4 ).

Numerical Pain Scale s : D eg flood analogue scale on 0 (I have no pain) to 10 (I have a pain in the degree intolerably) at the desired point is marked by giving a score between acquaint feel the pain severity of patients (5 ).

The parameters to be used in the research are used routinely.

ELIGIBILITY:
İnclusion criteria:

* Being between the ages of 18-60 who have previously been diagnosed with fibromyalgia
* Symptoms last longer than 3 months
* The volunteer's acceptance of participation in the treatment that will continue 2 days a week for 6 weeks

Exclusion criteria from the study:

* Using psychotropic medication in the last month
* Known central or peripheral nervous system disease, progressive neurological damage,
* Any serious cardiovascular pathology.
* Any musculoskeletal disease other than fibromyalgia,
* Presence of uncontrolled hypertension,

Exclusion criteria:

* Volunteer's request to leave
* Failure to continue training sessions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Short Form-36 | 6 weeks
  The Short Form-36 is a 36-item short-form questionnaire measuring eight health-related quality-of-life domains: physical functioning (PF), social functioning (SF), role limitation due to physical problems (RP), emotional problems (RE), mental health (MH), energy and vitality (VT), bodily pain (BP), and general health perception (GH). The SF-36 also includes an item for assessing changes in participant's health status over the past year. It is a scale between 0 (worst) and 100 (best) using the standard SF-36 scoring algorithms, with item scores coded, aggregated for each quality of life domain tested.
Fibromyalgia Impact Questionnaire | 6 weeks
  The Fibromyalgia Impact Questionnaire (FEA) measures 10 different characteristics: physical function, well-being, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. With the exception of the well-being trait, low scores indicate recovery or less affliction. FEA is filled by the patient. The maximum possible score of each sub-title is 10. Thus, the total maximum score is 100. The average FM patient scores 50, while more severely affected FM patients usually score above 70.
Numerical Pain Scale | 6 weeks
  Numerical Analog Scale (NAS) A scale with values from 0 to 10. Pain in the last 24 hours is evaluated with NAS. If 0 on the scale, I have no pain and 10 means unbearable pain and it is reported that the severity of the pain increases from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu Unıversity, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No